CLINICAL TRIAL: NCT06113185
Title: Turkish Psychometric Properties of Pain Behavior Scale in Patients With Chronic Low Back Pain
Brief Title: Psychometric Properties of Pain Scale in Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-15/518
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Chronic Low Back Pain
Keywords: Psychometric Properties; Pain Behavior Scale
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — Demographic and clinical information of the participants will be recorded using a standardized form. The cognitive status of the patient will be evaluated according to the answers to the questions asked to the patient during the questioning of demographic data and reading and signing the consent form. The participants will be asked to complete a series of questionnaires to assess pain intensity and characteristics, pain-related functional disability, and pain-related fear-avoidance behavior. To record the presence and severity of pain behaviors exhibited during physical performance tests, patients will be asked to complete 5 functional tests (repetitive trunk flexion, repetitive sit-to-stand, timed get-up-and-go test, reach with load, 50-step walk test) and observers will simultaneously complete the Pain Behavior Scale. Each participant will be asked to attend two testing sessions separated by one week and occurring before the start of treatment.

SUMMARY:
The aim of this study was to examine the Turkish validity of the Pain Behavior Scale in a population with chronic non-specific low back pain and to examine both intra-rater and inter-rater reliability. In addition, since this test package includes a series of functional activities, it is aimed to assess pain behaviors during functional movement in this population and to verify the test-retest reliability of physical performance tests.

DETAILED DESCRIPTION:
To assess the extent to which individuals with chronic low back pain are affected during functional task performance, the presence or absence of pain behaviors and the severity of observed pain behavior should be considered. The Pain Behavior Scale has potential clinical application both for assessing pain behaviors during regular physical examination and for measuring the presence and severity of pain behaviors during functional movement. There is no similar assessment tool that offers all of these simultaneously. Therefore, this study aimed to examine the Turkish validity of the Pain Behavior Scale in a population with chronic non-specific low back pain and to test its intra- and inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain for more than three months
* Being between the ages of 18-55
* Adequate cognitive functions (reading, writing, recall, orientation, language)

Exclusion Criteria:

* Presence of a serious underlying pathology (e.g. cancer, infection or cauda equina syndrome)
* Presence of spinal stenosis
* Presence of signs of radiculopathy (presence of neural symptoms such as pain radiating to the lower extremities, weakness, numbness and tingling sensation)
* Presence of fracture or surgical history in the relevant area
* Presence of rheumatic disease history
* Presence of pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients on the waiting list with a diagnosis of chronic nonspecific low back pain who applied to the Physical Therapy and Rehabilitation Outpatient Clinic of Acıbadem Health Group hospitals with complaints of low back pain will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Pain Behavior Scale | At the beginning of the study and up to 1 weeks
  The Pain Behavior Scale was developed to record the presence and severity of pain behaviors exhibited during physical performance tests. Specific pain behaviors assessed are sighing, breath holding, grimacing, guarding, rubbing and antalgic gait. The Pain Behavior Scale consists of a 4-point scale ranging from "None" (no observed behavior) to "Severe" (marked pain behavior).
  Two measures are obtained from the scale
  1. The presence or absence of each behavior
  2. Total score for the severity of general pain behaviors. The scale will be used during the implementation of physical performance tests lasting 10-15 minutes.
Visual Analog Scale | At the beginning of the study
  The Visual Analog Scale, which is used to record the intensity of pain, consists of a single 10 cm line; the left end is described as "No pain" and the right end is described as "The most severe pain experienced in life". Patients will be asked to mark the severity of their current pain on the 10 cm line. During the calculation, the marked point will be measured in cm. The higher the score, the more severe the pain.
McGill Pain Questionnaire-Short Form | At the beginning of the study
  The McGill Pain Questionnaire Short Form consists of three parts. In the first part, patients are asked to describe their pain with 15 descriptive words (11 sensory and 4 affective). In the second part, the severity of the patient's pain is evaluated. In the third part, patients are asked to mark their current pain intensity on a visual comparison scale.

SECONDARY OUTCOMES:
Oswestry Disability Index | At the beginning of the study
  The Oswestry Disability Index consists of 10 questions questioning the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleeping, the degree of change in pain, travel and social life and the questions are scored between 0-5. The total score is calculated as a percentage and the higher the total score, the higher the level of functional disability.
Fear-Avoidance Beliefs Questionnaire | At the beginning of the study
  The Fear-Avoidance Beliefs Questionnaire consists of two subscales, physical activity and work, and a total of 16 questions (5 physical activity sections and 11 work sections). The questionnaire is a 7-point Likert-type scale. In the answers to the questionnaire, 0 points are given for strongly disagree and 6 points are given for strongly agree. Both subscale scores can be used independently.

CONTACTS AND LOCATIONS:
Overall Officials: Elif E Safran, asst. prof., Principal Investigator — Acibadem Healthcare Group; Irmak Çavuşoğlu, asst. prof., Study Chair — Acibadem Healthcare Group; Nuray Alaca, assoc. prof., Study Director — Acibadem Healthcare Group
Locations (1):
- Acıbadem Health Group, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided